CLINICAL TRIAL: NCT03303365
Title: Cyberknife Radiosurgery for Patients With Brain Metastases Diagnosed With Either SPACE or MPRAGE Sequence - A Prospective Randomized Evaluation of Response and Toxicity
Brief Title: Cyberknife Radiosurgery for Patients With Brain Metastases Diagnosed With Either SPACE or MPRAGE Sequence
Acronym: CYBER-SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juergen Debus (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Prof. Dr.Dr. Jürgen Debus, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-448/2017
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Brain Metastases; Adult Solid Tumor
Keywords: Brain Metastases; WBRT (whole brain radiotherapy); SRS (stereotactic radiosurgery); CYBER-Knife
MeSH Terms: conditions — Brain Neoplasms; Snyder Robinson syndrome | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment based on SPACE MRI sequence (Experimental): Cyberknife SRS of all suspect intracranial lesions visible in SPACE up to 10 simultaneous lesions
  Interventions: Radiation: stereotactic radiosurgery (SRS)
- Treatment based on MPRAGE (Active Comparator): Cyberknife SRS of all suspect intracranial lesions visible in MPRAGE up to 10 simultaneous lesions
  Interventions: Radiation: stereotactic radiosurgery (SRS)

INTERVENTIONS:
Radiation: stereotactic radiosurgery (SRS) — All patients will receive a pre-treatment cranial MRI for diagnostic and treatment planning purposes.
  In Arm A, the contrast-based T1-weighted SPACE sequence is utilized for GTV definition. In Arm B, the contrast-based T1-weighted three-dimensional MPRAGE sequence is utilized for GTV definition. In both cases the GTV consists of all contrasted tissue associated with the target lesion and all additional tissue judged by an experienced physician to be part of the suspect target lesion. To the GTV a PTV margin of 1 mm is added by isotropic expansion that can be slightly modified if deemed necessary by the treating physician (e.g. intersection with adjoining OAR).
  Dose prescription to the PTV for target lesions will be as follows:
  * 20 Gy to the 70%-isodose (lesions < 2 cm max. diameter)
  * 18 Gy to the 70%-isodose (lesions 2 - 3 cm max. diameter)
  * 6 x 5 Gy to the conformally surrounding isodose (lesions > 3 cm max. diameter)

SUMMARY:
For patients with cerebral oligometastases who are in adequate clinical condition stereotactic radiosurgery (SRS) is the treatment of choice, being recommended by international guidelines for the treatment of one to four lesions. Newer findings have shown that for patients with more than four lesions SRS can be considered as a favorable alternative to whole-brain radiotherapy (WBRT), the currently established standard-of-care treatment. With modern techniques highly conformal SRS of multiple lesions has become feasible with comparable clinical effort and minimal toxicity as compared to WBRT. Developments in magnetic resonance imaging (MRI- imaging) have produced highly sensitive contrast-enhanced three-dimensional fast spin echo sequences such as SPACE that facilitate the detection of very small and early-stage lesions in a fashion superior to the established Magnetization Prepared Rapid Gradient Echo (MPRAGE) series.

Since it has been established that the response of brain metastases to SRS is better for smaller lesions and that WBRT can come at the price of significant neurotoxicity, the investigators hypothesize that 1) earlier detection of small brain metastases and 2) early and aggressive treatment of those by SRS will result in an overall clinical benefit by delaying the failure of repeated localized therapy and thus preserving quality of life and potentially prolonging overall survival. On the other hand however, overtreatment might be a valid concern with this approach since it has yet to be proved that a clinical benefit can be achieved.

The current study aims to stretch the boundaries of the term "cerebral oligometastases" by performing SRS for up to ten cerebral metastases, compared to the established clinical standard of four, given that existing data supports the non-inferiority of this approach and given that modern Cyberknife SRS facilitates the treatment of multiple lesions with minimal treatment-associated toxicity.

DETAILED DESCRIPTION:
Scientific Background: Brain metastases are the most common intracranial cancer manifestations, affecting up to one third of adult cancer patients with systemic spread. Prognosis is generally poor with overall survival ranging below 6 months on average. However, a more detailed inspection reveals a prognostic subgroup, for which improved overall survival and clinical symptom control can be achieved and that is most descriptively characterized by favorable clinical performance (KPI ≥ 70%) and extracranially controlled disease. Whereas for most patients with brain metastases whole-brain radiotherapy, steroids or best supportive care represent the palliation treatment of choice, the abovementioned subgroup is eligible to profit from a locally radical therapy concept and in those cases neurosurgical resection and stereotactic radiosurgery have both produced favorable results. In patients unsuitable for neurosurgical resection, single- or multifraction, SRS has several distinct advantages over WBRT, the most significant being short treatment time, less posttherapeutic neurocognitive impairment, better local tumor control and little to no hair loss. Furthermore, SRS can be repeated multiple times or performed before or after WBRT. Current clinical guidelines recommend SRS in cases of cerebral oligometastases, defined as one to four intracranial lesions with an extracranially controlled systemic disease status. However, recent data suggests that it may be a suitable treatment for patients with five to ten or even more than ten lesions, being non-inferior to the SRS of four or less lesions. There are several factors supporting this rationale: On the one hand technical improvements in the field of SRS have significantly facilitated the treatment of a higher number of target lesions with little to no increase in toxicity and comparable clinical effort. On the other hand, the ever improving sensitivity of medical imaging has caused an increase in the detection of oligometastatic constellations, enabling their treatment in an earlier stage. For a long time the contrast-based high-resolution cranial computer tomography (cCT) had been the gold standard of detecting cerebral metastases. This was significantly improved by the introduction of magnetic resonance imaging (MRI) with contrast-enhanced T1-weighted sequences. Sensitivity was further improved with the introduction of 3T MRI into clinical routine and the development of high-resolution three-dimensional gradient-echo sequences such as the contrast-based T1-weighted MPRAGE, featuring a slice thickness of 0.9 mm and multiplanar reconstruction, thus enabling the detection of very small sized lesions in the range of one to a few millimeters. However, the use of gradient-echo (GE) techniques to obtain three-dimensional high-spatial-resolution images comes at the cost of inferior contrast enhancement and higher susceptibility to artifacts than is the case with two-dimensional spin-echo (SE) techniques. Recent developments in MRI research have produced another sequence that might prove even superior to MPRAGE in the specific detection of very small and early brain metastases: Sampling perfection with application-optimized contrasts by using different flip angle evolutions (SPACE) is a three-dimensional fast SE sequence that combines high contrast enhancement superior to MPRAGE with a high spatial resolution and multiplanar reconstruction. Kato et al. have found this sequence to be significantly superior to MPRAGE in the detection of contrast enhanced parenchymal lesions, especially if those are < 5mm in size as is characteristic of small very-early-stage cerebral metastases.

Trial Objectives: It is the purpose of this study to evaluate treatment response and toxicity after SRS of up to ten simultaneous cerebral metastases, treating either all lesions visible in the highly sensitive SPACE MRI sequence or only those visible in the conventional contrast-based MPRAGE sequence. Treatment response is evaluated with respect to the ineligibility for further cerebral SRS at 12 months after initial SRS, defined by simultaneous new occurrence or progression of > 10 brain metastases (as a surrogate parameter for overall local control), furthermore overall survival and cognitive function and quality of life.

Patients´Selection: A total of n=200 patients will be enrolled into the trial (n=100 per treatment group). All patients fulfilling the inclusion and exclusion criteria will be informed about the study and included into the study if they declare informed consent. Registration for the study must be performed before the start of RT.

Trial Design: The trial will be performed as a single-center two-armed prospective randomized Phase II study. Patients will be randomized into an experimental arm and a control arm. All patients will receive pre-therapeutic MRI imaging as described in (Chapter 6) and imaging will be assessed by a radiologist. For patients in the experimental arm, all available MRI series, including SPACE will be taken into consideration for the definition of treatment target lesions. For patients in the control arm the assessing radiologist will be blinded with respect to the SPACE sequence and for the definition of treatment target lesions primarily contrast-based three-dimensional MPRAGE, complemented by all non-SPACE MRI sequences will be taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* radiologically confirmed metastases of the brain with an underlying history of a malignant illness
* between one and ten suspect intracranial lesions, taking into consideration all available series of the pre-therapeutic MRI (performed at Heidelberg University Hospital and including SPACE sequence)
* age ≥ 18 years of age
* Karnofsky Performance Score (KPS) ≥ 70
* for women with childbearing potential, (and men) adequate contraception.
* ability to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patient to take part in the study
* Small-cell lung cancer (SCLC) as primary malignant illness
* More than 10 suspect intracranial lesions in the initial pre-therapeutic MRI imaging (performed at Heidelberg University Hospital and including SPACE sequence)
* metastasis so close to OAR that initial single-session SRS would be impossible due to lacking radiotolerance
* known contraindications against the performing of cranial MRI
* previous radiotherapy of the brain
* Patients who have not yet recovered from acute toxicities of prior therapies
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Ineligibility for further cerebral SRS | 12 months after initial SRS
  simultaneous new occurrence or progression of > 10 brain metastases

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months after initial SRS
  Time interval between the date of RT begin and the date of death or date of leaving the study e.g., lost to follow up) whatever occurs first.
cognitive function | 6 months after initial SRS
  CANTAB Test (Cambridge Neuropsychological Test Automated Battery )
quality of life | 6 months after initial SRS
  EORTC QLQ-C30 questionnaire to assess the QoL of cancer patients, clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof. Dr.Dr., Principal Investigator — Head of department Radiation Oncology
Locations (1):
- University Hospital of Heidelberg, Department of Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson JD, Young B. Demographics of brain metastasis. Neurosurg Clin N Am. 1996 Jul;7(3):337-44. PMID 8823767
- [Background] Arvold ND, Lee EQ, Mehta MP, Margolin K, Alexander BM, Lin NU, Anders CK, Soffietti R, Camidge DR, Vogelbaum MA, Dunn IF, Wen PY. Updates in the management of brain metastases. Neuro Oncol. 2016 Aug;18(8):1043-65. doi: 10.1093/neuonc/now127. PMID 27382120
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Sperduto PW, Berkey B, Gaspar LE, Mehta M, Curran W. A new prognostic index and comparison to three other indices for patients with brain metastases: an analysis of 1,960 patients in the RTOG database. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):510-4. doi: 10.1016/j.ijrobp.2007.06.074. Epub 2007 Oct 10. PMID 17931798
- [Background] Linskey ME, Andrews DW, Asher AL, Burri SH, Kondziolka D, Robinson PD, Ammirati M, Cobbs CS, Gaspar LE, Loeffler JS, McDermott M, Mehta MP, Mikkelsen T, Olson JJ, Paleologos NA, Patchell RA, Ryken TC, Kalkanis SN. The role of stereotactic radiosurgery in the management of patients with newly diagnosed brain metastases: a systematic review and evidence-based clinical practice guideline. J Neurooncol. 2010 Jan;96(1):45-68. doi: 10.1007/s11060-009-0073-4. Epub 2009 Dec 4. PMID 19960227
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Wowra B, Muacevic A, Tonn JC. CyberKnife radiosurgery for brain metastases. Prog Neurol Surg. 2012;25:201-9. doi: 10.1159/000331193. Epub 2012 Jan 6. PMID 22236681
- [Background] Mugler JP 3rd, Bao S, Mulkern RV, Guttmann CR, Robertson RL, Jolesz FA, Brookeman JR. Optimized single-slab three-dimensional spin-echo MR imaging of the brain. Radiology. 2000 Sep;216(3):891-9. doi: 10.1148/radiology.216.3.r00au46891. PMID 10966728
- [Background] Kato Y, Higano S, Tamura H, Mugikura S, Umetsu A, Murata T, Takahashi S. Usefulness of contrast-enhanced T1-weighted sampling perfection with application-optimized contrasts by using different flip angle evolutions in detection of small brain metastasis at 3T MR imaging: comparison with magnetization-prepared rapid acquisition of gradient echo imaging. AJNR Am J Neuroradiol. 2009 May;30(5):923-9. doi: 10.3174/ajnr.A1506. Epub 2009 Feb 12. PMID 19213825
- [Background] Mulkern RV, Wong ST, Winalski C, Jolesz FA. Contrast manipulation and artifact assessment of 2D and 3D RARE sequences. Magn Reson Imaging. 1990;8(5):557-66. doi: 10.1016/0730-725x(90)90132-l. PMID 2082125
- [Background] Kakeda S, Korogi Y, Hiai Y, Ohnari N, Moriya J, Kamada K, Hanamiya M, Sato T, Kitajima M. Detection of brain metastasis at 3T: comparison among SE, IR-FSE and 3D-GRE sequences. Eur Radiol. 2007 Sep;17(9):2345-51. doi: 10.1007/s00330-007-0599-9. Epub 2007 Feb 22. PMID 17318603
- [Background] Chang EL, Hassenbusch SJ 3rd, Shiu AS, Lang FF, Allen PK, Sawaya R, Maor MH. The role of tumor size in the radiosurgical management of patients with ambiguous brain metastases. Neurosurgery. 2003 Aug;53(2):272-80; discussion 280-1. doi: 10.1227/01.neu.0000073546.61154.9a. PMID 12925241
- [Background] Aoyama H, Tago M, Kato N, Toyoda T, Kenjyo M, Hirota S, Shioura H, Inomata T, Kunieda E, Hayakawa K, Nakagawa K, Kobashi G, Shirato H. Neurocognitive function of patients with brain metastasis who received either whole brain radiotherapy plus stereotactic radiosurgery or radiosurgery alone. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1388-95. doi: 10.1016/j.ijrobp.2007.03.048. PMID 17674975
- [Background] Chang SD, Main W, Martin DP, Gibbs IC, Heilbrun MP. An analysis of the accuracy of the CyberKnife: a robotic frameless stereotactic radiosurgical system. Neurosurgery. 2003 Jan;52(1):140-6; discussion 146-7. doi: 10.1097/00006123-200301000-00018. PMID 12493111
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Shultz DB, Modlin LA, Jayachandran P, Von Eyben R, Gibbs IC, Choi CYH, Chang SD, Harsh GR 4th, Li G, Adler JR, Hancock SL, Soltys SG. Repeat Courses of Stereotactic Radiosurgery (SRS), Deferring Whole-Brain Irradiation, for New Brain Metastases After Initial SRS. Int J Radiat Oncol Biol Phys. 2015 Aug 1;92(5):993-999. doi: 10.1016/j.ijrobp.2015.04.036. Epub 2015 Apr 28. PMID 26194677
- [Background] Shen CJ, Rigamonti D, Redmond KJ, Kummerlowe MN, Lim M, Kleinberg LR. The strategy of repeat stereotactic radiosurgery without whole brain radiation treatment for new brain metastases: Outcomes and implications for follow-up monitoring. Pract Radiat Oncol. 2016 Nov-Dec;6(6):409-416. doi: 10.1016/j.prro.2016.04.004. Epub 2016 Apr 26. PMID 27687187
- [Background] van Buuren S. Multiple imputation of discrete and continuous data by fully conditional specification. Stat Methods Med Res. 2007 Jun;16(3):219-42. doi: 10.1177/0962280206074463. PMID 17621469
- [Background] Higgins JP, White IR, Wood AM. Imputation methods for missing outcome data in meta-analysis of clinical trials. Clin Trials. 2008;5(3):225-39. doi: 10.1177/1740774508091600. PMID 18559412